CLINICAL TRIAL: NCT02199340
Title: The iStep Study: Development and Validation of an Incremental Exercise Step Test for Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11AR14
Record Dates: First submitted 2014-06-12; First posted 2014-07-24 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
Keywords: Exercise testing; Children; Exercise capacity
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cystic fibrosis (Experimental): * iStep exercise test
  * CPET exercise test
  Interventions: Other: iStep exercise test; Other: CPET exercise test
- Healthy control (Active Comparator): - iStep exercise test
  Interventions: Other: iStep exercise test

INTERVENTIONS:
Other: iStep exercise test — newly developed submaximal exercise test
Other: CPET exercise test — maximal gold standard exercise test
  Arms: Cystic fibrosis

SUMMARY:
The progression of lung disease in cystic fibrosis (CF) results inevitably in a reduction in exercise capacity. The assessment of fitness and exercise capacity in CF is an important measure of the impact of the disease process, particularly if it is repeated over time. With recent advances in clinical management, CF lung disease in children can be relatively mild and exercise tolerance good. The currently available field tests e.g. 3 minute step test, are often completed too easily. These tests provide limited information relating to maximal exercise performance. By contrast, the maximal CardioPulmonary Exercise Test (CPET), a progressive, incremental, gold standard exercise test with breath by breath analysis of expired gas, has proved to be a valuable means of assessing exercise response in patients with CF. Its only limitation is the requirement for specialist laboratory facilities, equipment and staff.

A new field test for evaluating exercise capacity in children is needed. This should be portable, easy to administer and simple to perform by young children, while providing a higher intensity of exercise which correlates with day to day activity patterns of children, and clinically relevant information in the short term and longitudinally. This test needs to be a good surrogate measure of exercise capacity when formal CPET is unable to be undertaken. By providing accurate and useful information the results can be used to prescribe and train individuals with CF safely and effectively and can also be used in the short and long term for guidance of the medical management of these complex patients.

The aim of this study is to develop and validate the use of a new incremental step test to assess exercise tolerance/capacity in children with CF, compare this with the gold standard CPET and to provide normative healthy control comparison data The main objectives of the study are

1. To develop an incremental step test to assess exercise tolerance / capacity in children with CF.
2. To compare the incremental step test with the gold standard CPET
3. To assess the level of exercise response produced by the incremental step test
4. To assess the correlation between independent variables of lung function measurements, age, weight and height with VO2peak and other exercise test outcomes
5. To assess the repeatability and evaluate the normal variability of the new incremental step test
6. To provide healthy control normative data for comparison

ELIGIBILITY:
Inclusion Criteria:

Clinical population inclusion

* Parental/guardian consent
* Participant assent
* Male or female
* Confirmed Cystic fibrosis diagnosis (by genetic genotype or positive sweat test)
* Receiving physiotherapy as part of their usual care
* Height >125cm to allow cycle ergometer use
* 6-16 years

Healthy control population inclusion

* Parental/guardian consent
* Participant assent
* Male or female
* 6-16 years

Exclusion Criteria:

Clinical population exclusion

* <6 years and >16 years
* No consent / assent
* Frank haemoptysis in the last 48 hours
* Acute infective exacerbation (defined as increased temperature, additional antibiotics)
* Poor dietary intake/hydration
* Oxygen dependent at rest
* Arterial oxygen saturation (SaO2) <90% at rest
* Burkholderia cepacia
* Coexisting insulin dependent diabetes mellitus
* Methicillin-resistant Staphylococcus aureus (MRSA) positive

Healthy control population exclusion

* <6 years and >16 years
* No consent / assent
* Acute infection (defined as increased temperature and antibiotics)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) | Measured during the exercise test, day 1, maximum of 20 minutes
  Gold standard exercise test to determine peak oxygen uptake during exercise

SECONDARY OUTCOMES:
Secondary breath by breath analysis outcome measures | Measured during the exercise test, day 1, maximum of 20 minutes
Newly developed iStep exercise test outcome variables | Measured during the exercise test, day 1, maximum of 20 minutes
  Standard field exercise test outcomes of heart rate, oxygen saturations, time, level achieved, rate of perceived exertion, perceived breathlessness
Height, weight and body mass index measures | Measured at baseline on the day of testing, day 1, maximum of 5 minutes
  Height, weight and body mass index will be measured for descriptive purposes only
Reasons for termination of the incremental step test | Measured at the end of the exercise test, day 1, maximum of 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rand, BA, BSc, MSc, Principal Investigator — UCL Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided